CLINICAL TRIAL: NCT03536572
Title: Self-Management of Continuous Positive Airway Pressure Settings for Veterans With Sleep Apnea
Brief Title: Self-Management of Continuous Positive Airway Pressure Settings
Acronym: ImPRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IIR 16-277
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Sleep Apnea Syndromes; Chronic Disease; Adherence; Self-Care; Patient Outcomes
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Chronic Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep Apnea Self-Management Program (Active Comparator): Protocol-based sleep apnea and CPAP education and support
  Interventions: Behavioral: Sleep Apnea Self-Management Program
- Individualized Pressure Adjustment (Experimental): Additional education and support that will allow them to adjust their PAP pressures
  Interventions: Behavioral: Sleep Apnea Self-Management Program

INTERVENTIONS:
Behavioral: Sleep Apnea Self-Management Program — Protocol-based sleep apnea and CPAP education and support
  Other Names: SASMP

SUMMARY:
Obstructive sleep apnea (OSA) is a major chronic condition affecting the quality of life of millions of Americans. Per the Institute of Medicine new treatment adherence strategies are needed to help improve the quality of care, reduce social and economic costs, and help those with chronic conditions, including OSA, live healthier and more productive lives through better management of their conditions. Adherence with continuous positive airway pressure (PAP) therapy is disappointingly low, and new methods to increase both the use and efficacy of therapy are needed. Historically, patients have not been formally instructed to adjust their pressure settings on their PAP devices; practically, however, allowing patients to adjust their pressure settings fosters engagement, self-confidence, and control with therapy.

DETAILED DESCRIPTION:
Because of clinical demands, patients are often under-educated and under-supported about the features of their positive airway pressure (PAP) devices. The most engaged patients are ones who understand the details of their device and change the feature settings so that they can maximize the benefits of therapy. Features settings include humidification level, expiratory pressure relief, pressure ramping, mask alert, auto pressure start, among other important comfort features. Historically, patients have not been provided with access to alter or modify therapy pressure settings, which requires physician prescription. Allied medical staff can carry out subsequent pressure setting changes. It is clear that it is difficult for the healthcare system to engage in optimal chronic disease management, and accommodate the needs of sleep apnea patients early in the treatment initialization process, which requires multiple visits/contacts to ensure that patients are maximizing the use of therapy.

The overarching aim of the proposed project is to examine the effect of providing patients with the ability to adjust their PAP pressure levels on therapy adherence and outcomes. To answer these research questions, the proposed randomized, controlled two-group trial of Sleep Apnea Self-Management Program (SM) and SM plus Individualized Pressure Adjustment (IPA) has the following specific aims related to APAP adherence and efficacy, patient-reported outcomes, and utilization: (1) To examine the effect of Individualized Pressure Adjustment (IPA) of settings on treatment adherence and efficacy (i.e., mask leak and residual apnea-hypopnea index); (2) To examine the effect of SM+IPA versus SM on patient self-reported treatment outcomes; and (3) To describe the effects of SM-IPA and SM groups on utilization.

Sleep apnea is one of the most common chronic conditions in the VA. Positive airway pressure (PAP) therapy is the gold-standard therapy for sleep apnea, but adherence with PAP is suboptimal. VA sleep programs are understaffed relative to clinical demand for education and support. While adaption to PAP therapy has traditionally been achieved through sequential visits and pressure changes initiated by providers during office-based care, self-monitoring and individualized pressure adjustment is an important strategy that would empower Veterans to achieve better control of their OSA. The key impacts of this project are significant for both patients (improved outcomes) and the VA (improved staff efficiencies).

While patients have control over a wide range of comfort features on their PAP devices, historically they have not been formally educated and supported to adjust pressure settings. The unique aspect of this study is the focus on individualizing pressure settings to allow for the maximizing therapeutic benefit, including increased PAP adherence. Importantly, this is done within the context of provider oversight.

The proposed study is a 6-month randomized, controlled, non-blinded, single-center study comparing the Sleep Apnea Self-Management Program (SM) to SM plus Individualized Pressure Adjustment (IPA). Both groups will receive the SM protocol to ensure that they receive identical OSA and PAP education and support. Participants in the intervention arm will be provided with additional education and support that will allow them to adjust their PAP pressures.

Positive findings from this study will result in a Toolkit that can be distributed to provide patients and providers with the knowledge necessary to improve the clinical management of OSA.

ELIGIBILITY:
Inclusion Criteria:

The investigators' intent is to recruit a study population that is representative of patients diagnosed with OSA. To this end, entry criteria are as inclusive as possible and operationalized as follows:

* confirmed diagnosis of OSA
* being newly prescribed an OSA therapy
* having chronic symptoms per screening symptom checklist
* fluency in English
* receiving medical care at VA San Diego Healthcare System

OSA diagnosis by the investigators' Pulmonary Sleep Program has been and is currently consistent with published consensus statements50 that therapy is indicated when the apnea-hypopnea index (AHI, number of apneas + hypopneas per hour of sleep) is either (1) >30 or (2) 5-30 AND accompanied by documented OSA symptoms, including EDS, impaired cognition, mood disorders, insomnia, or documented cardiovascular diseases. Because sleep apnea is of increasing importance in women, the investigators' plan is to oversample women by 50% so that they represent 15% of the final study sample.

Exclusion Criteria:

Criteria for exclusion include:

* cognitive impairment sufficient to cause inability to complete the protocol (e.g., documented MMSE < 24/30)
* low health literacy
* residence in a geographical area outside of San Diego County (which could make some necessary in-person visits difficult)
* fatal comorbidity (life expectancy <6 months as indicated by treating physician)
* significant documented substance/chemical abuse
* other participant circumstances or characteristics that, in the opinion of a consensus of study team, would interfere with the safety of a prospective participant or their need for treatment (i.e.,:)

  * clinical needs of patient outweighs needs of research study

No exclusion criteria or any other study design elements will be used directly or indirectly to restrict study participation by women or members of minority groups. Some minority groups are thought to have higher OSA prevalence rates than Caucasians, so assuming they are being screened/diagnosed at the same rates as Caucasians, the investigators expect minority groups to be included in the study at levels equal to or higher than the VA San Diego minority composition.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl J Stepnowsky, Jr., PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sleep Apnea Self-Management Program | Individualized Pressure Adjustment
Started | 134 | 136
Completed | 96 | 113
Not Completed | 38 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sleep Apnea Self-Management Program | Individualized Pressure Adjustment | Total
Number analyzed (Participants) | 96 | 113 | 209
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 90 | 104 | 194
  >=65 years | 6 | 9 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (11.8) | 48.1 (12.6) | 47.27 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 83 | 105 | 188
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 14 | 26 | 40
  Native Hawaiian or Other Pacific Islander | 2 | 4 | 6
  Black or African American | 21 | 15 | 36
  White | 54 | 62 | 116
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 96 | 113 | 209
Apnea-Hypopnea Index [Mean (Standard Deviation); unit: Events per hour] — The AHI is measured on a numeric scale. Scores for adults are divided into three categories, which correspond to different levels of OSA severity. The AHI range is from 0 to ~140. It is true there is no upper true maximum, but above 140 is extremely unlikely:
  Normal: An AHI between 0 and fewer than 5. Mild: An AHI of at least 5 events per hour, but fewer than 15. Moderate: An AHI of at least 15 events per hour, but fewer than 30. Severe: An AHI of at least 30 events per hour.
  Events per hour | 24.5 (21.6) | 26.3 (23.2) | 25.5 (22.4)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Adherence
Description: Measurement of the amount of time that CPAP is used on average per night over the outcome time frame
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: Hours per night
Arm/Group | Sleep Apnea Self-Management Program | Individualized Pressure Adjustment
Number analyzed (Participants) | 96 | 113
Hours per night | 2.1 (1.5) | 2.2 (1.6)

ADVERSE EVENTS:
Time Frame: 1 month and 2 months.
Arm/Group | Sleep Apnea Self-Management Program | Individualized Pressure Adjustment
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/113
Other Adverse Events (participants affected / at risk) | 0/96 | 0/113

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT03536572/Prot_SAP_000.pdf